CLINICAL TRIAL: NCT02692651
Title: A Comparison of Fidaxomicin and Oral Vancomycin for the Treatment of Clostridium Difficile Infection (CDI) in Hospitalized Patients Receiving Concomitant Antibiotics for the Treatment of Concurrent Systemic Infections
Brief Title: A Comparison of Fidaxomicin and Vancomycin in Patients With CDI Receiving Antibiotics for Concurrent Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Krishna Rao, Assistant Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Merck Fidaxo
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Results first posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Clostridium Difficile Infection (CDI)
Keywords: vancomycin; fidaxomicin; CDI; diarrhea
MeSH Terms: conditions — Clostridium Infections; Diarrhea | interventions — Fidaxomicin; OPT 80; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fidaxomicin (Active Comparator): Fidaxomicin 200 mg PO BID for 10 days or until the end of the duration of concomitant antibiotic exposure, whichever is longer.
  Interventions: Drug: Fidaxomicin
- Vancomycin (Active Comparator): Vancomycin 125 mg PO QID for 10 days or until the end of the duration of concomitant antibiotic exposure, whichever is longer.
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Fidaxomicin — Eligible patients randomized to receive open-label Fidaxomicin will receive 200 mg twice daily for 10 days or until the end of the duration of concomitant antibiotics exposure, whichever is longer.
  Other Names: Dificid, Dificlir, OPT-80, PAR-101
  Arms: Fidaxomicin
Drug: Vancomycin — Eligible patients randomized to Vancomycin will receive 125 mg orally four times daily for 10 days or until the end of the duration of concomitant antibiotics exposure, whichever is longer.
  Other Names: Vancocin
  Arms: Vancomycin

SUMMARY:
Administration of concomitant antibiotics (CA) is a known risk factor for treatment failure in the treatment of CDI, as well as for recurrence of CDI. Recent data suggested that among patients receiving CA, fidaxomicin is superior to vancomycin. While these data are encouraging, many clinicians remain unclear on how to apply these data to patient care. Additionally, patients were excluded from the trials presented to the FDA if it was expected that they would require ≥ 7 days of CA. Therefore, the clinical question still remains of how to apply these data to the real world patient who requires a long course of CA and develops CDI while on therapy. We therefore propose an open label, comparative and prospective study of fidaxomicin 200 mg twice daily vs oral vancomycin 125 mg four times daily for the treatment of CDI among patients who are receiving a long course of CA.

We hypothesize that fidaxomicin will be superior to vancomycin with respect to clinical cure for patients with CDI.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older with >3 unformed stools/24 hours with positive stool test for C. difficile.
* Patients receiving ≥ 1 high or medium risk antibiotic for treatment of an infection other than CDI, for an anticipated duration of ≥ 5 days from the time of enrollment.

  * High risk: carbapenems, 2nd-4th generation cephalosporins, fluoroquinolones, clindamycin, and beta-lactam/beta-lactamase inhibitor combinations
  * Medium risk: 1st generation cephalosporin, macrolides*, and aztreonam

    * *The macrolide would be considered to be low risk if patients are receiving intermittent macrolides for prophylaxis only and not for treatment of an acute infection

Exclusion Criteria:

* Patients with severe-complicated disease that would compromise oral therapy (hypotenstion or shock, ileus or bowel obstruction, megacolon).
* Patients with an allergy to oral vancomycin or fidaxomicin.
* Patients anticipated to receive metronidazole after enrollment.
* Patients who already received oral vancomycin or metronidazole (either oral or intravenous) for > 24 hours within the preceding 72 hours at the time of enrollment.
* Patients anticipated to receive adjunctive C. difficile therapy (rifaxamin, nitazoxanide, tigecycline) after enrollment.
* Patients who are on laxatives before they are enrolled into the study, such as lactulose, if:

  * Patients have had a recent dose adjustment;
  * Baseline number of bowel movement while on laxatives is unknown.
  * Number of bowel movements and/or consistency has not changed from baseline.
* Patients who have had colostomy or ileostomy
* Patients who will have colostomy or ileostomy after enrollment and before study ends
* Patients who are or will be on long-term (>12 weeks) medium or high-risk antibiotics prophylaxis after enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-05-23 (Actual); Study Completion 2021-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Krishna Rao, MD, MS, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - St. Joseph Mercy Hospital, Ypsilanti, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rao K, Zhao Q, Bell J, Krishnan J, Henig O, Daniel J, Sawaya K, Albin O, Mills JP, Petty LA, Gregg K, Kaul D, Malani AN, Pogue J, Kaye KS. An Open-Label, Randomized Trial Comparing Fidaxomicin With Oral Vancomycin for the Treatment of Clostridioides difficile Infection in Hospitalized Patients Receiving Concomitant Antibiotics for Concurrent Infections. Clin Infect Dis. 2024 Feb 17;78(2):277-282. doi: 10.1093/cid/ciad606. PMID 37797310

RESULTS

PARTICIPANT FLOW:
Groups:
- Vancomycin: Vancomycin solution 125 mg PO 4 times per day for 10 days or until the end of the duration of concomitant antibiotic exposure, whichever is longer.
- Fidaxomicin: Fidaxomicin pill 200 mg PO 2 times per day for 10 days or until the end of the duration of concomitant antibiotic exposure, whichever is longer.
Period: Study Treatment
Arm/Group | Vancomycin | Fidaxomicin
Started | 70 | 74
Completed | 54 | 64
Not Completed | 16 | 10
Not completed — Death | 7 | 3
Not completed — comfort care | 1 | 1
Not completed — Protocol violation per treating team preference | 8 | 6
Period: Post Study Treatment Follow-up
Arm/Group | Vancomycin | Fidaxomicin
Started | 54 | 64
Completed | 50 | 60
Not Completed | 4 | 4
Not completed — Death | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fidaxomicin | Vancomycin | Total
Number analyzed (Participants) | 74 | 70 | 144
Age, Customized [Count of Participants; unit: Participants]
  <65 | 51 | 40 | 91
  65-74 | 15 | 20 | 35
  >74 | 8 | 10 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 35 | 75
  Male | 34 | 35 | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 5 | 15
  White | 61 | 61 | 122
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 74 | 70 | 144
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 26.7 [15.5 to 48.2] | 28.2 [15.2 to 51.3] | 27.4 [15.2 to 51.3]
Patients in ICU at enrollment [Count of Participants; unit: Participants] — Number of patients who were in the Intensive Care Unit (ICU) when enrolled.
  Participants | 12 | 11 | 23
History of C difficile infection [Count of Participants; unit: Participants] | 16 | 8 | 24
History of cancer [Count of Participants; unit: Participants] | 34 | 38 | 72
History of stem cell transplant [Count of Participants; unit: Participants] | 4 | 10 | 14
History of inflammatory bowel disease [Count of Participants; unit: Participants] | 3 | 2 | 5
History of Proton Pump Inhibitors use [Count of Participants; unit: Participants] | 29 | 30 | 59
White blood cell count [Mean (Full Range); unit: 1000 cells/μL] | 9.46 [0.1 to 33.5] | 7.93 [0.1 to 36.3] | 8.7 [0.1 to 36.3]
Creatinine [Mean (Full Range); unit: mg/dl] | 1.11 [0.26 to 3.27] | 1.36 [0.42 to 5.36] | 1.23 [0.26 to 5.36]

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure: Resolution of Diarrhea
Description: Resolution of diarrhea defined as ≤ 3 unformed stools for 2 consecutive days maintained until the end of therapy and for 2 days afterwards. The treatment course was at least 10 days, but it could be extended to a maximum of 12 weeks.
Time Frame: length of treatment plus 2 days, from a minimum of 12 to a maximum of 86 days
Population: Intention to treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 74 | 70
Participants | 54 | 44
Statistical Analysis 1: Comparison: Fidaxomicin vs Vancomycin; Test type: Superiority; p = 0.195, Chi-squared, Corrected

2. Secondary Outcome: Recurrence of CDI
Description: Recurrence is defined as all three of the following within 4 weeks after successfully completing study treatment: reappearance of symptoms of CDI (>3 unformed stools in a 24 hour period; a positive stool PCR test for C. difficile; and the need for retreatment with an agent active against C. difficile).
Time Frame: 30 days after treatment's end (maximum of 114 days)
Population: Subjects who completed study treatment and were alive at the end of 30-day follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 60 | 50
Participants | 2 | 2
Statistical Analysis 1: Comparison: Fidaxomicin vs Vancomycin; Test type: Superiority; p = .99, Chi-squared, Corrected

3. Secondary Outcome: 30-day Mortality
Description: Death in subjects who completed the study treatment and died within 30 days after end of treatment
Time Frame: 40 to 114 days
Population: Subjects who completed the study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 64 | 54
Participants | 4 | 4
Statistical Analysis 1: Comparison: Fidaxomicin vs Vancomycin; Test type: Superiority; p = .999, Chi-squared, Corrected

ADVERSE EVENTS:
Time Frame: Treatment period + 30 days, ranging from a total of 40 to 114 days.
Description: Adverse events collected with follow-up surveys and by clinical alerts.
Arm/Group | Fidaxomicin | Vancomycin
All-Cause Mortality (participants affected / at risk) | 7/74 | 11/70
Serious Adverse Events (participants affected / at risk) | 11/74 | 13/70
Other Adverse Events (participants affected / at risk) | 0/74 | 0/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fidaxomicin (N=74) | Vancomycin (N=70)
Hospitalization (Gastrointestinal disorders) | 5 (5) | 2 (2)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 4 (4)
Hospitalization (Infections and infestations) | 0 (0) | 4 (4)
Hospitalization (Renal and urinary disorders) | 1 (1) | 1 (1)
Hospitalization (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hospitalization (Nervous system disorders) | 1 (1) | 2 (3)
Hospitalization (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Hospitalization (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT02692651/Prot_SAP_000.pdf